CLINICAL TRIAL: NCT01679808
Title: Pressure Dependent Tracheal Obstruction in Copd Patients
Acronym: PDTO
Status: Completed | Type: Observational
Sponsor: LHL Helse (Other)
Responsible Party: Sponsor
Other Study IDs: GK-18; s-04058c (Registry Identifier: The National Committees for Research Ethics in Norway)
Record Dates: First submitted 2012-09-03; First posted 2012-09-06 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2012-09

CONDITIONS: Tracheobronchomalacia
Keywords: copd; airway obstruction; Tracheobronchomalacia
MeSH Terms: conditions — Tracheobronchomalacia; Pulmonary Disease, Chronic Obstructive; Airway Obstruction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Background. Do pressure dependent tracheal obstructions (PDTO) often seen during bronchoscopy in COPD patients affect pulmonary function tests and breathing symptoms? Method. Model study. A garden hose was compressed from one side to simulate the posterior wall of the trachea bulging into the lumen. For two obstruction lengths - 3 cm and 12 cm, the hose was increasingly compressed in eight steps. Resistance was measured at each step for airflows 1 l/s through 9 l/s, and digital photos of the luminal area were taken which were used by a computer to estimate the cross sectional area reduction and the corresponding distance between the bulging (posterior)and the opposite (anterior) wall (AP-distance).

Patient study. 104 stable COPD patients studied by pulmonary function tests and bronchoscopy. The tracheal obstruction was observed during forced expiration and cough, and the cross sectional area reduction was estimated using the results from the model study.

ELIGIBILITY:
Inclusion Criteria:

* copd

Exclusion Criteria:

* clinical evidence of malignant disease
* not able to be subjected to bronchoscopy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients (both sexes) in a pulmonary rehabilitation clinic
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2004-08; Primary Completion 2006-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivar Ellingsen, Dr med, Principal Investigator — LHL Helse
Locations (1):
- Glittreklinikken, Hakadal, Akershus, Norway